CLINICAL TRIAL: NCT01280162
Title: An Active Malaria Epidemiology Cohort Study With Evaluation of a 2 Day Versus 3 Day Treatment Regimen of Dihydroartemisinin (DHA)-Piperaquine for Patients With Uncomplicated Malaria
Brief Title: Malaria Active Epidemiology and Treatment Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Armed Forces Research Institute of Medical Sciences, Thailand (Other Government)
Collaborators: United States Army Medical Materiel Development Activity (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WRAIR # 1737; HRPO Log Number A-16251 (Registry Identifier: US Army Medical Research and Materiel Command)
Record Dates: First submitted 2011-01-19; First posted 2011-01-20 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Malaria
Keywords: Plasmodium falciparum, Plasmodium vivax
MeSH Terms: conditions — Malaria; Malaria, Falciparum; Malaria, Vivax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3 day therapy (Experimental): Total dose split over 3 days (3 tablets per day)
  Interventions: Drug: Dihydroartemisinin piperaquine
- 2 day therapy (Experimental): Total dose split over 2 days (4.5 tablets per day)
  Interventions: Drug: Dihydroartemisinin piperaquine

INTERVENTIONS:
Drug: Dihydroartemisinin piperaquine — 40/320 mg tablets, 9 tablets total
  Other Names: Artekin, Duo-cotexcin

SUMMARY:
An observational cohort and malaria treatment study in Cambodia.

DETAILED DESCRIPTION:
This is an active observational Cohort Study of malaria epidemiology with a nested two arm, randomized, open label Treatment Study comparing the efficacy, safety, tolerability and pharmacokinetics of a two versus three day course of Dihydroartemisinin-Piperaquine (DP) for those developing uncomplicated malaria. At the conclusion of the Cohort Study, a subset of volunteers with documented exposure to Plasmodium vivax during the study will be treated with primaquine as presumptive anti-relapse therapy directed against the exoerythrocytic malaria stages of P. vivax, and followed passively for an additional 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Otherwise healthy volunteer, 18-65 years of age, eligible for care at an RCAF facility, and at risk for contracting malaria
2. Able to provide informed consent
3. Likely to reside in endemic area for the duration of the study
4. Available for follow-up for anticipated study duration, and agrees to participate for the duration of the study
5. Authorized by local commander to participate in the study if on active duty

Exclusion Criteria:

1. History of allergic reaction or contraindication to DHA or piperaquine
2. Significant acute comorbidity requiring urgent medical intervention
3. Pregnant or lactating female, or a female of childbearing age who does not agree to use a highly effective method of birth control during the study
4. Clinically significant abnormal EKG, including a QTc interval > 500 ms.
5. Judged by the investigator to be otherwise unsuitable for study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2010-09; Primary Completion 2011-02 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Adequate clinical and parasitological response to a treatment regimen of DHA-PIP for Plasmodium falciparum | 6 months
  Number of malaria recurrences for 2 and 3 day DHA-PIP drug regimens within 42 days after treatment of malaria infection, diagnosed by positive PCR-corrected malaria microscopy.

SECONDARY OUTCOMES:
Number of Cambodian study subjects with reduced or null activity hepatic cytochrome P450 2D6 alleles | 1 year
  Using Polymerase Chain Reaction-based bead array assays, genotype the human hepatic CYP2D6 allele in study participants giving informed consent for genetic testing
Number of subjects with reduced or null hepatic CYP2D6 enzyme phenotype using activity-score A system | 1 year
  For each CYP2D6 genotype determined, use the AS-A system to assign predicted metabolism phenotype

CONTACTS AND LOCATIONS:
Overall Officials: Michele D. Spring, MD, MSPH, Principal Investigator — USAMC-AFRIMS
Locations (1):
- Oddar Meancheay, Anlong Veaeng, Cambodia

REFERENCES:
- [Background] Lon C, Manning JE, Vanachayangkul P, So M, Sea D, Se Y, Gosi P, Lanteri C, Chaorattanakawee S, Sriwichai S, Chann S, Kuntawunginn W, Buathong N, Nou S, Walsh DS, Tyner SD, Juliano JJ, Lin J, Spring M, Bethell D, Kaewkungwal J, Tang D, Chuor CM, Satharath P, Saunders D. Efficacy of two versus three-day regimens of dihydroartemisinin-piperaquine for uncomplicated malaria in military personnel in northern Cambodia: an open-label randomized trial. PLoS One. 2014 Mar 25;9(3):e93138. doi: 10.1371/journal.pone.0093138. eCollection 2014. PMID 24667662
- [Derived] Vanachayangkul P, Lon C, Spring M, Sok S, Ta-Aksorn W, Kodchakorn C, Pann ST, Chann S, Ittiverakul M, Sriwichai S, Buathong N, Kuntawunginn W, So M, Youdaline T, Milner E, Wojnarski M, Lanteri C, Manning J, Prom S, Haigney M, Cantilena L, Saunders D. Piperaquine Population Pharmacokinetics and Cardiac Safety in Cambodia. Antimicrob Agents Chemother. 2017 Apr 24;61(5):e02000-16. doi: 10.1128/AAC.02000-16. Print 2017 May. PMID 28193647
- [Derived] Spring MD, Pichyangkul S, Lon C, Gosi P, Yongvanichit K, Srichairatanakul U, Limsalakpeth A, Chaisatit C, Chann S, Sriwichai S, Auayapon M, Chaorattanakawee S, Dutta S, Prom S, Meng Chour C, Walsh DS, Angov E, Saunders DL. Antibody profiles to plasmodium merozoite surface protein-1 in Cambodian adults during an active surveillance cohort with nested treatment study. Malar J. 2016 Jan 8;15:17. doi: 10.1186/s12936-015-1058-8. PMID 26747132
- [Derived] Spring MD, Lin JT, Manning JE, Vanachayangkul P, Somethy S, Bun R, Se Y, Chann S, Ittiverakul M, Sia-ngam P, Kuntawunginn W, Arsanok M, Buathong N, Chaorattanakawee S, Gosi P, Ta-aksorn W, Chanarat N, Sundrakes S, Kong N, Heng TK, Nou S, Teja-isavadharm P, Pichyangkul S, Phann ST, Balasubramanian S, Juliano JJ, Meshnick SR, Chour CM, Prom S, Lanteri CA, Lon C, Saunders DL. Dihydroartemisinin-piperaquine failure associated with a triple mutant including kelch13 C580Y in Cambodia: an observational cohort study. Lancet Infect Dis. 2015 Jun;15(6):683-91. doi: 10.1016/S1473-3099(15)70049-6. Epub 2015 Apr 12. PMID 25877962
- See also: Publication describing results of clinical trial — https://journals.plos.org/plosone/article?id=10.1371/journal.pone.0093138
- See also: Publication describing CYP2D6 alleles in this Cambodian study population — https://www.ajtmh.org/content/journals/10.4269/ajtmh.20-0061